CLINICAL TRIAL: NCT05928702
Title: The Effect of Temperature-elevating Armbaths (Hauffe-Schwenniger-Baths) as a Therapeutic Option to Regulate the Blood Pressure in People With Arterial Hypertension - a Randomized-controlled Trial (Wirksamkeit Temperaturansteigender Armbäder (Hauffe-Schweninger Bäder) Zur Regulierung Des Blutdrucks Bei Probanden Mit Arterieller Hypertonie - Eine Randomisiert-kontrollierte Studie)
Brief Title: Temperature-elevating Armbaths for Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Kohl, Wiebke, MD, Kliniken Essen-Mitte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WKHypertension
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Arterial Hypertension
Keywords: Complementary Medicine; Hydrotherapy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Armbath (Experimental): The armbath group will perform a temperature-elevating armbath developed by Hauffe and Schwenninger. A large bowl and a thermometer will be given to each participant.
  Participant start with bathing their forearms up to about one third of the upper arm in a large bowl with water at approximately 37°C. Within 30min, they are advised to add hot water to the bowl for multiple times until a temperature of 42°C. After 30min, the arms can be taken out of the water, dried, and participants are recommended to rest for additional 30 min afterwards.
  Prior medication should be continued throughout the whole trial.
  Interventions: Procedure: temperature-elevating armbath
- Waitlist (No Intervention): Participants will continue their treatment as usual (e.g. medication). After the end of the trial (6 months) they will be offered to get instructed on performing temperature-elevating armbaths.

INTERVENTIONS:
Procedure: temperature-elevating armbath — Hydrotherapeutic Approach
  Arms: Armbath

SUMMARY:
The goal of this randomized controlled trial is to learn about the effect of a hydrotherapeutic approach - a temperature-elevating armbath - in people with arterial hypertention. The main question[s] it aims to answer are:

* Can this kind of hydrotherapy lower the blood pressure and therefore be an additional approach to medical treatment in arterial hypertension?
* Besides blood pressure regulation, does this intervention affect sleep quality when being performed at night time or does it affect overall quality of life?

Participants will be advised to perform a temperature-elevating armbath once a day for 30 minutes on at least 5 days per week over 8 weeks.

The comparison group will continue treatment as usual, like continue their medication. 24h blood pressure measurements will be performed at the beginning, after 8 weeks and after 6 months in both groups. The main goal is to evaluate whether the intervention group shows lower blood pressure levels after a certain time of treatment.

After 6 months (end of trial) the control group will be offered to learn the temperature elevating armbath as well.

DETAILED DESCRIPTION:
Arterial hypertension remains one of the most important risk factors in developing a cardiovascular disease. While medical treatment is usually necessary, lifestyle modifications should always be included. Besides physical activity and a balanced diet, there are also therapeutic approaches from the so called classical complementary medicine. One very important part in Europe is hydrotherapy, based on ideas of Sebastian Kneipp and his contemporaries. In hydrotherapy there are various therapeutic approaches that can be used additionally to conventional therapy. Because conventional medical therapy is often associated with unwanted side effects, these additional approaches experience increasing popularity. In arterial hypertension, temperature-elevating armbaths, developed by Kneipps contemporaries Hauffe and Schwenninger, are a hydrotherapeutic approach that is highly recommended. Even though hydrotherapy has been a part of complementary medicine for more than a century now some therapeutic approaches lack of scientific evidence - especially when it comes to their effect on arterial hypertension.

This randomized-controlled trial aims to evaluate the effect of a temperature-elevating armbath among participants with arterial hypertension. 50 participants will be randomized to either an intervention group or waitlist (treatment as usual). All 50 participants will be monitored with three 24-hours ambulatory blood pressure measurements (24h ABPM) at the beginning of the trial after randomization, at 8 weeks and at 6 months.

The intervention group will be advised to perform the armbaths on 5 of 7 days per week for 8 weeks total. Each participant will get a detailed instruction how to perform the armbath and will be handed a diary to document their performance.

After 6 months, each participant of the control group will be offered to be instructed on performing the armbaths as well.

Within the active period of 8 weeks, participants of both groups will be called regularly to ask about their health and whether they have questions regarding the trial.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (≥18 years)
* diagnosed arterial hypertension, at least stage I, based on the Guidelines of the European Society of Hypertension 2018 (systolic >140 mmHg, diastolic >90 mmHg)
* last change in medication at least 2 months ago
* no planned changes in blood pressure medication within intervention time; changes due to medical reasons (e.g., hypotension, hypertensive emergency) are allowed.
* willingness to perform an armbath on a regular schedule (min. 5x/weeks)

Exclusion Criteria:

* acute psychiatric disease ( e.g., addiction, major depression)
* acute or major physical disease (e.g., cancer diagnosis within the last 5 years, major known cardiovascular diseases, renal or liver dysfunction), acute infection, major neurological diseases (e.g., Parkinsons´ disease, uncontrolled epilepsy)
* secondary hypertension
* pregnancy or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | to 8 weeks

SECONDARY OUTCOMES:
Blood pressure | to 6 months
SF-12 | to 8 weeks and 6 months
  Health-related quality of life
PSQI | to 8 weeks and 6 months
  Sleep quality
heartrate | to 8 weeks and 6 months
Adverse events | to 8 weeks and 6 months
Medication | to 8 weeks and 6 months
  Monitoring of changes in medication

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Blood pressure measurements, Comorbidities, medication